CLINICAL TRIAL: NCT03118297
Title: Intervention to End Recurrent Unscheduled Bleeding Trial: A Randomized-controlled Trial of Ulipristal Acetate for Unscheduled Bleeding in Etonogestrel Implant Users
Brief Title: Intervention to End Recurrent Unscheduled Bleeding Trial
Acronym: INTERRUPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rachel Zigler, MD MSCI, Clinical Fellow, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201612002
Record Dates: First submitted 2017-04-04; First posted 2017-04-18 (Actual); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Contraception; Bleeding
Keywords: Etonogestrel Implant
MeSH Terms: conditions — Hemorrhage | interventions — ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ulipristal Acetate (Experimental): 15mg ulipristal acetate (capsule) daily for 7 days
  Interventions: Drug: Ulipristal Acetate
- Placebo (Placebo Comparator): Identical placebo (capsule) daily for 7 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Ulipristal Acetate — Women who have bothersome bleeding with the etonogestrel implant will be randomized to receive ulipristal acetate versus placebo daily for 7 days.
  Arms: Ulipristal Acetate
Drug: Placebo oral capsule — Women who have bothersome bleeding with the etonogestrel implant will be randomized to receive ulipristal acetate versus placebo daily for 7 days.
  Arms: Placebo

SUMMARY:
The subdermal etonogestrel (ENG) implant, a long-acting reversible contraceptive (LARC) method, is among the most effective forms of reversible contraception and thus, an important tool in the quest to reduce unintended pregnancy. However, despite overall increases in LARC use in the United States from 1.5% in 2002 to 7.2% in 2011, and 11.6% most recently in 2015, implant use continues to make up a small proportion of LARC use. While evidence to explain this low uptake of implants is lacking, one potential reason is patient and provider concerns about unpredictable bleeding.

As a result of this, many studies have been performed in attempts to discover therapies for unscheduled bleeding in progestin-only contraceptive users. Some of these studies include those investigating selective progesterone receptor modulators, such as mifepristone and ulipristal acetate (UPA), which did find some benefit. Although a previous study showed mixed benefit, the investigators feel that this medication has demonstrated both biologic plausibility as well as clinically important outcomes. This previous study may not be entirely translatable to the proposed research as therapies were used for different indications (prophylaxis vs. treatment) and different progestins and delivery systems were studied. Therefore, the investigators believe UPA should not be discounted as a potential therapy. UPA may provide an additional safe and effective option for treatment of irregular bleeding with implants in women. In addition, UPA is currently available in outpatient pharmacies in the U.S. as a single 30mg oral tablet.

The investigators propose to investigate UPA for the treatment of unscheduled and troublesome bleeding in ENG implant users.

DETAILED DESCRIPTION:
The subdermal etonogestrel (ENG) implant, a long-acting reversible contraceptive (LARC) method, is among the most effective forms of reversible contraception and thus, an important tool in the quest to reduce unintended pregnancy. Despite this, ENG implant users make up a small percent of overall women that use LARC in the United States. Previous studies have demonstrated that among women dissatisfied with their implant, the majority cite unpredictable and irregular bleeding as a primary reason. Dissatisfaction with a contraceptive method can lead to discontinuation, which can put a woman at risk for unplanned pregnancy. Although irregular bleeding is a common side effect of all progestin-only contraceptives, there are significant gaps in our knowledge regarding the etiology of and effective therapies for unscheduled bleeding. While several mechanisms have been proposed and therapies have been studied, lack of convincing scientific evidence, in addition to possible contraindications to these therapies, demonstrates the need to investigate additional effective interventions.

Studies evaluating interventions for abnormal uterine bleeding resulting from uterine leiomyoma provide insight into potential therapies for progestin-mediated bleeding. In prior studies, ulipristal acetate (UPA) has been shown to reduce bleeding symptoms associated with uterine leiomyoma, including decreasing or stopping excessive bleeding. Progestin-associated irregular bleeding has been proposed to be secondary to a disruption in endometrial angiogenesis, therefore creating a fragile venous network. UPA may displace local progestin to counteract this effect. Thus, this medication has demonstrated both biologic plausibility as well as clinically important benefits. UPA may provide an additional safe and effective option for treatment of irregular bleeding in implant users. As women are often dissatisfied with irregular bleeding with the implant as noted above, improving bleeding profiles could potentially improve uptake and continuation of the device.

The investigators will perform a double blinded, randomized, placebo-controlled trial. Women will be randomized to receive either 15mg of UPA daily for 7 days or placebo for the same duration. The investigators hypothesize that UPA will decrease bleeding and spotting days in users of the ENG implant with unscheduled bleeding when compared to placebo as assessed by daily bleeding diaries.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-45
* Implant placed >90 days and <3 years prior to enrollment
* Patient complaint of bothersome irregular bleeding with implant
* Willing to be abstinent or use condoms during study period
* Willing to complete 30-day bleeding diary
* Willing to be randomized to placebo or ulipristal acetate
* Ability to send/receive SMS text message

Exclusion Criteria:

* Non-English speaking
* Implant placed >3 years prior to enrollment
* Contraindication to ulipristal acetate (current use of barbiturates, bosentan, carbamazepine, felbamate, griseofulvin, oxcarbazepine, phenytoin, rifampin, St. John's Wort, topiramate, known or suspected pregnancy, hypersensitivity to active substance or excipients, uterine/cervical/ovarian/breast cancer, severe asthma insufficiently controlled by oral glucocorticoids)
* Inability or unwillingness to comply with medication protocol
* Inability or unwillingness to comply with bleeding diary
* Breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Zigler, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zigler RE, Madden T, Ashby C, Wan L, McNicholas C. Ulipristal Acetate for Unscheduled Bleeding in Etonogestrel Implant Users: A Randomized Controlled Trial. Obstet Gynecol. 2018 Oct;132(4):888-894. doi: 10.1097/AOG.0000000000002810. PMID 30130351

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Identical appearing placebo (capsule) daily for 7 days
  Placebo oral capsule: Women who have bothersome bleeding with the etonogestrel implant will be randomized to receive ulipristal acetate versus placebo daily for 7 days.
Period: Overall Study
Arm/Group | Ulipristal Acetate | Placebo
Started | 32 | 33
Completed | 32 | 31
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ulipristal Acetate | Placebo | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants lost to follow up in placebo group
  years
    number analyzed (Participants) | 32 | 31 | 63
    (all) | 26.4 (6.2) | 25.5 (6.3) | 26.0 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants lost to follow up in placebo group
  Participants
    number analyzed (Participants) | 32 | 31 | 63
    Female | 32 | 31 | 63
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 participants lost to follow up in placebo group
  Participants
    number analyzed (Participants) | 32 | 31 | 63
    Hispanic or Latino | 0 | 2 | 2
    Not Hispanic or Latino | 32 | 29 | 61
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 2 participants lost to follow up in placebo group
  Participants
    Race: number analyzed (Participants) | 32 | 31 | 63
    Race: Black | 20 | 21 | 41
    Race: White | 7 | 7 | 14
    Race: Other or multiracial | 5 | 3 | 8
Region of Enrollment [Number; unit: participants] — Population: 2 participants lost to follow up in placebo group
  participants
    United States: number analyzed (Participants) | 32 | 31 | 63
    United States | 32 | 31 | 63
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: 2 participants lost to follow up in placebo group
  kg/m^2
    number analyzed (Participants) | 32 | 31 | 63
    (all) | 29.6 (8.2) | 27.8 (7.0) | 28.7 (7.6)
Duration of implant use [Median (Inter-Quartile Range); unit: months] — Population: 2 participants lost to follow up in placebo group
  months
    number analyzed (Participants) | 32 | 31 | 63
    (all) | 10.9 [5.5 to 18.1] | 9.2 [5.9 to 19.3] | 10.1 [5.7 to 18.7]
Days of bleeding in 30 days prior to enrollment [Median (Inter-Quartile Range); unit: days] — Population: 2 participants lost to follow up in placebo group
  days
    number analyzed (Participants) | 32 | 31 | 63
    (all) | 20.5 [12.5 to 29.5] | 20.0 [14.0 to 28.0] | 20.3 [13.3 to 28.8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding/Spotting Days With Use of Ulipristal Acetate as Measured by Daily Bleeding Diaries
Description: To evaluate the effectiveness of ulipristal acetate (15mg) in decreasing bleeding/spotting days due to the ENG implant over a 30-day period as compared to placebo.
Time Frame: 30 days
Population: See baseline characteristics
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ulipristal Acetate | Placebo
Number analyzed (Participants) | 32 | 31
days | 7 [4.5 to 11.0] | 12 [6.0 to 21.0]
Statistical Analysis 1: Comparison: Ulipristal Acetate vs Placebo; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney) — Threshold for significance: p=0.05

2. Secondary Outcome: Number of Participants With Bleeding Cessation by Day 10
Description: To evaluate bleeding cessation rates by day 10 following seven days of treatment with either ulipristal acetate or placebo.
Time Frame: 10 days
Population: See baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ulipristal Acetate | Placebo
Number analyzed (Participants) | 32 | 31
Participants | 11 | 3
Statistical Analysis 1: Comparison: Ulipristal Acetate vs Placebo; Test type: Superiority; p = 0.032, Fisher Exact — Threshold for significance: p=0.05

3. Secondary Outcome: Participant Satisfaction With Bleeding Pattern at 30 Days
Description: To evaluate participant satisfaction with regards to bleeding pattern after use of ulipristal acetate.
Time Frame: 30 days
Population: See baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ulipristal Acetate | Placebo
Number analyzed (Participants) | 32 | 31
Participants
  Not at all happy | 0 | 7
  Somewhat unhappy | 0 | 2
  Neither happy nor unhappy | 4 | 3
  Somewhat happy | 5 | 10
  Very happy | 23 | 8
  Did not respond | 0 | 1
Statistical Analysis 1: Comparison: Ulipristal Acetate vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Threshold for significance: p=0.05

4. Secondary Outcome: Number of Participants With Medication Side Effects by 30 Days
Description: To evaluate participant satisfaction with regards to medication side effects.
Time Frame: 30 days
Population: See baseline characteristics
Measure: Number; unit: participants
Arm/Group | Ulipristal Acetate | Placebo
Number analyzed (Participants) | 32 | 31
participants
  Headache | 3 | 6
  Nausea/Vomiting | 1 | 3
  Feeling flushed | 0 | 1
  Abdominal pain | 2 | 2
  Dizziness | 1 | 1
  Other | 1 | 1
  Did not experience | 26 | 23
Statistical Analysis 1: Comparison: Ulipristal Acetate vs Placebo; Test type: Superiority; p > 0.05, Chi-squared — Threshold for significance: p=0.05

5. Secondary Outcome: Ovulation Status Measured by Weekly Serum Progesterone Levels
Description: To evaluate effect, if any, of ulipristal acetate on ovulation status. Data in the table represent the lowest and highest values that were recorded over all of the measurements for each arm as a whole.
Time Frame: Baseline, weeks 1, 2, 3, 4
Population: See baseline characteristics
Measure: Number; unit: ng/mL
Arm/Group | Ulipristal Acetate | Placebo
Number analyzed (Participants) | 32 | 31
ng/mL
  Lower endpoint | 0.0 | 0.0
  Upper endpoint | 4.4 | 1.3
Statistical Analysis 1: Comparison: Ulipristal Acetate vs Placebo; Test type: Other — No statistical test performed; Significance testing not performed. All values below prespecified limit of 5.0 ng/mL

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ulipristal Acetate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT03118297/Prot_SAP_000.pdf